CLINICAL TRIAL: NCT04263285
Title: Treatment of Depression Post-SCI: Retrospective Analysis and Feasibility Trial
Brief Title: Treatment of Depression Post-SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Catherine VanDerwerker, Research Associate, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00086228
Record Dates: First submitted 2020-02-04; First posted 2020-02-10 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Depression; Spinal Cord Injuries
MeSH Terms: conditions — Depression; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- rTMS (Repetitive Transcranial Magnetic Stimulation) (Experimental)
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — The study team will deliver rTMS five days a week for four weeks, according to a specific and approved protocol for participant positioning, motor threshold determination, and dosing.

SUMMARY:
Depression is more common after a spinal cord injury (SCI) than in the general population. Unfortunately, it is unknown how depression is typically treated in individuals with SCI or if commonly used treatment methods are effective. This study will investigate the safety and impact of a novel method for treating depression called repetitive transcranial magnetic stimulation (rTMS). rTMS is a type of non-invasive brain stimulation. Fourteen individuals with a cervical or thoracic level SCI and depression will complete an approved treatment plan using rTMS. Participants will be treated using rTMS five days a week for four weeks. After four weeks of treatment, the study team will review the safety of rTMS and assess changes in depressive symptoms. If the results are positive, larger studies can be designed to develop better treatment options for individuals with SCI and depression.

ELIGIBILITY:
Inclusion criteria:

1. Age 18 - 70;
2. At least 6 months post incomplete cervical or incomplete or complete thoracic level SCI;
3. Have at least partial active movement of the right thumb (abductor pollicis brevis) to allow for FDA approved rTMS dosing;
4. Major depressive disorder, as identified through screening tools;
5. No antidepressant medications or no change in doses of psychotropic medication(s) for at least 4 weeks prior to the study (6 weeks if newly initiated medication).

Exclusion criteria:

1. Concomitant neurologic diseases/disorders or dementia;
2. Cognitive impairment, as identified through a screening tool (Montreal Cognitive Assessment);
3. History of major head trauma as identified through a screening tool (Ohio State University Traumatic Brain Injury Identification Method);
4. History of psychosis or other Axis I disorder that is primary;
5. Positive screen for bipolar disorder, as identified through a screening tool (The Mood Disorder Questionnaire);
6. Life expectancy <1 year;
7. Attempt of suicide in the last 2 years;
8. Electronic or metallic implants (i.e. metal in the head, cochlear implant, or pacemaker);
9. History of seizures or currently prescribed anti-seizure medications;
10. Taking medication that increases the risk of seizures;
11. Pregnancy as identified through a positive pregnancy test;
12. Inability or unwillingness of subject or legal guardian/representative to give informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by number of adverse events | Through the study period (5 weeks)
  Report of adverse and serious adverse events in all participants.
Number of visits missed | Throughout the treatment period (4 weeks)
  The average of the number of intervention visits missed across all participants
Change in depressive symptoms as assessed by the Hamilton Rating Scale for Depression | Baseline, midpoint (Week 3), and post treatment (5 weeks)
  The Hamilton Rating Scale for Depression consists of 17 questions with a total score range from 0 - 52. Ranges of total score include the following: 0 - 7 suggests normal/no depressive symptoms; 8 - 16 suggests mild depressive symptoms; 17 - 23 suggests moderate depressive symptoms; and 24 - 52 suggests severe depressive symptoms.

SECONDARY OUTCOMES:
Change in depressive symptoms as assessed by the Montgomery- Asberg Depression Rating Scale (MADRS) | Baseline, midpoint (Week 3), and post treatment (5 weeks)
  Montgomery- Asberg Depression Rating Scale consists of 10 questions with a range of 0 - 60.
  Ranges of total score include the following: 0 - 6 suggest normal/ no depressive symptoms; 7 - 19 suggests mild depressive symptoms; 20 - 34 suggests moderate depressive symptoms; and 34 - 60 suggests severe depressive symptoms.
Change in the impact depressive symptoms have on one's life as assessed by the Sheehan Disability Scale. | Baseline, midpoint (Week 3), and post treatment (5 weeks)
  The Sheehan Disability Scale is a self-report questionnaire that assess how depressive symptoms have impacted one's ability to participate in work/school, social life, and family life. Each question is scored from 0 (not at all) to 10 (extremely). Total score ranges from 0 (unimpaired) to 30 (highly impaired).
Change in subjective well-being based on the Satisfaction With Life Scale. | Baseline and post treatment (5 weeks)
  The Satisfaction With Life Scale is a self-report questionnaire regarding subjective well-being. The scale consists of 5 questions that are rated between 1 (Strongly Disagree) to 7 (Strongly Agree). Pre and post intervention answers will be compared.
Change in physical activity based on the Leisure Time Physical Activity Questionnaire for People with Spinal Cord Injury | Baseline and post treatment (5 weeks)
  Self-report questionnaire regarding the number of days and minutes an individual participates in mild, moderate, and heavy intensity physical activity/effort. Pre and post intervention answers will be compared.
Change in function as assessed by the Spinal Cord Independence Measure III-Self Report. | Baseline and post treatment (5 weeks)
  The Spinal Cord Independence Measure III-Self Report is a self-report questionnaire regarding the degree of assistance needed for daily self care activities, such as eating, bathing, dressing, grooming, breathing, bladder and bowel management, toileting, transfers, and mobility. There are a total of 17 questions with a total score of 0 (assistance required) to 100 (no assistance or mobility aids). Pre and post intervention scores will be compared.
Change in function and daily activities as assessed by the Craig Handicap Assessment and Reporting Tool-Short Form | Baseline and post treatment (5 weeks)
  The Craig Handicap Assessment and Reporting Tool-Short Form is a self-report questionnaire that includes a total of 19 questions regarding physical assistance, cognitive assistance, mobility, occupation, social integration, and financial resources. Pre and post intervention answers will be compared.
Change depressive symptoms as assessed by the Patient Health Questionnaire-9 score | Baseline, midpoint (Week 3), and post treatment (5 weeks)
  The Patient Health Questionnaire-9 is a 9 questions self-report measure of depressive symptoms. The total score ranges from 0 - 27. Ranges of total score include the following: 0 suggests no depressive symptoms; 1 - 4 suggests minimal depressive symptoms; 5 - 9 suggests mild depressive symptoms; 10 - 14 suggests moderate depressive symptoms;15 - 19 suggests moderately severe depressive symptoms; and 20 - 27 suggests severe depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine VanDerwerker, DPT, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No